CLINICAL TRIAL: NCT02470533
Title: Transarterial Chemoembolization With Drug-Eluting Beads (Standard Arm) Versus Stereotactic Body Radiation Therapy (Experimental Arm) for Hepatocellular Carcinoma: A Multicenter Randomized Phase II Trial
Brief Title: Transarterial Chemoembolization Versus Stereotactic Body Radiation Therapy for Hepatocellular Carcinoma
Acronym: TRENDY
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Erasmus Medical Center (Other)
Collaborators: Dutch Cancer Society (Other); UMC Utrecht (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); VU University of Amsterdam (Other); Radboud University Medical Center (Other); Maastricht University Medical Center (Other); Maastro Clinic, The Netherlands (Other); Leiden University Medical Center (Other); Universitaire Ziekenhuizen KU Leuven (Other); University Hospital, Antwerp (Other); University Hospital, Lille (Other)
Responsible Party: Principal Investigator, Alejandra Mendez Romero, MD PhD, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL51318.078.14
Record Dates: First submitted 2015-06-08; First posted 2015-06-12 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Liver Neoplasms
MeSH Terms: conditions — Liver Neoplasms | interventions — Radiotherapy; Chemoembolization, Therapeutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transarterial chemoembolization (Active Comparator): Chemoembolization will be performed through a transarterial route delivering drug eluting beads, i.e. hydrogel-based microspheres (Biocompatibles UK, Ltd, HepaSphere Biosphere Medical) loaded with the chemotherapeutic agent doxorubicin.
  Interventions: Device: chemoembolization
- Stereotactic body radiation therapy (Experimental): Risk-adapted dose prescription for delivering the highest possible tumor dose not exceeding the maximum dose in 6 fractions of 8-9 Gy, while hepatic normal tissue complication probability (NTCP) < of 5%
  Interventions: Radiation: Radiation therapy

INTERVENTIONS:
Radiation: Radiation therapy — 6 fractions of 8-9Gy
  Arms: Stereotactic body radiation therapy
Device: chemoembolization — Up to 4 sessions
  Arms: Transarterial chemoembolization

SUMMARY:
Rationale:

This study will compare head to head in patients with hepatocellular carcinoma (HCC) ineligible for surgery or radiofrequency ablation, the standard treatment arm, transarterial chemoembolization with drug-eluting beads (TACE-DEB), with the experimental arm, stereotactic body radiation therapy (SBRT). The investigators hypothesis is that the time to progression is more favorable after SBRT than after TACE-DEB. The expected time to include the required patients for this trial will be four years.

To the best of the investigators knowledge this study will be the first in the world that will compare both techniques in a randomized trial.

Objective:

To assess the time to progression after TACE-DEB and after SBRT in a comparable population of patients diagnosed with HCC.

Study design:

Randomized, prospective, open-label, and phase II study.

Study population:

Patients diagnosed with HCC, Child-Pugh grade A, one to three tumors, cumulative diameter ≤ 6cm, and ≥ 18 years old.

Intervention:

Patients with HCC will be randomized to receive the standard treatment, TACE-DEB loaded with doxorubicin or the experimental arm, SBRT.

Main study parameters/endpoints:

The primary endpoint of this study will be time to progression, defined as time from randomization to radiological progression.

Secondary endpoints will be:

* Time to local recurrence
* Response rate (complete and partial response)
* Overall survival
* Toxicity
* Quality of life.

DETAILED DESCRIPTION:
Primary liver cancer, particularly hepatocellular carcinoma (HCC) is a major health problem. Curative therapies for HCC are considered hepatic resection, liver transplantation and radiofrequency ablation (RFA). Hepatic resection is preferred for patients with limited disease, non-cirrhotic livers or selected patients with Child-Pugh A cirrhosis. Unlike resection, liver transplantation treats the tumor and the underlying cirrhosis present in the liver. Candidates for liver transplantation are preferably those with cirrhosis and tumors that comply with the Milan criteria (single tumor <5cm or 1-3 tumors each of ≤ 3cm). Because most patients are not amenable to resection or liver transplantation, RFA has emerged as an effective treatment option. RFA is limited by the location of the tumor in the liver and by the tumor size with best results after RFA achieved for tumors ≤3cm. For patients that are not eligible for RFA due to large or multifocal tumors, transarterial chemoembolization with drug-eluting beads (TACE-DEB) is the preferred treatment.

Stereotactic body radiation therapy (SBRT) delivers a highly effective dose of irradiation to the tumor while maximally avoiding dose delivery to surrounding healthy structures. SBRT is offered as an ablative local treatment with reported high percentages of complete and partial responses with limited toxicity.

An international expert committee on HCC has recommended time to progression (TTP) as primary endpoint for phase II randomized trials. Although data is scarce the best published median TTP after TACE-DEB was 16 months and after SBRT 36.5months in a more or less comparable patient population (Barcelona Clinic Liver Cancer stage system A-C).

The present study will include patients not eligible for resection or RFA. Patients may be eligible for bridging or for down staging to transplantation. Well compensated liver cirrhosis (Child-Pugh A) and disease confined to the liver (one to three tumors cumulative diameter ≤ 6cm) is required. To our knowledge this trial will be the first in the world to compare TACE-DEB and SBRT. This trial may have a big impact on the control of the disease and may contribute to change the standard of care from a palliative to a more radical/curative intention in this patient population

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with HCC Patients can be included if they require treatment prior to liver transplantation.
* Barcelona Clinic Liver Cancer Stage System class A-B
* One to three tumors of maximum cumulative diameter ≤ 6 cm measured in all 3 axes.
* Measurable disease to be selected as a target on CT/MRI-scan, according to mRECIST criteria for HCC within 6 weeks prior to randomization (≥ 1cm at least in one dimension, suitable for repeated measurement, and arterial enhancement) [44].
* Tumor visibility on CT
* Child-Pugh A cirrhosis
* Age ≥ 18 years
* ECOG performance status 0-1
* Albumin> 28 g/l, bilirubin < 50 µmol/l, INR < 2.3, AST/ALT < 5 times ULN, within 6 weeks prior to randomization
* Platelets will be preferably ≥ 50x10E9/ l (if not, thrombocytes transfusion is allowed to ensure a safe procedure at the discretion of the interventional radiologist and gastroenterologist). Leukocytes > 1.5x10E9/l, Hb > 6 mmol/l, within 6 weeks prior to randomization
* Written informed consent
* Willing and able to comply to the follow-up schedule
* Planned to start treatment within 6 weeks from randomization.

Exclusion Criteria:

* Eligibility for resection or RFA
* More than three tumors in the liver
* Ascites
* Any signs of acute viral or non-viral hepatitis
* Encephalopathy
* Vascular tumor invasion (contact with the vessel will not be considered contraindication).
* Previous radiotherapy to the liver
* Known current pregnancy
* Distance from the tumor to the esophagus, stomach, duodenum, small bowel or large bowel < 0.5 cm on CT or on MRI (randomization imaging). Depending on the SBRT technique used, the minimum acceptable distance may vary and be larger for one technique compared to the other
* Uncontrolled portal hypertension (high bleeding risk). If gastroscopy has been performed, untreated esophageal varices grade III or IV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-04-30 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Time to progression | 4 years

SECONDARY OUTCOMES:
Time to local recurrence | 4 years
Response rate | 4 years
Overall survival | 4 years
Toxicity | 4 years
  Common toxicity criteria v4.0
Quality of life | 4 years
  EORTC Quality of life forms C-30 and HCC-18, Quality of life form Euro QoL5D

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra Mendez Romero, MD PhD, Principal Investigator — Erasmus Medical Center; Adriaan Moelker, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (11):
- Belgium (2):
  - UH Antwerp, Antwerp
  - UH Leuven, Leuven
- UH Lille, Lille, France
- Netherlands (8):
  - Erasmus MC, Rotterdam, South Holland
  - AMC, Amsterdam
  - VU MC, Amsterdam
  - LUMC, Leiden
  - Maastro, Maastricht
  - UMC Maastricht, Maastricht
  - UMC St Radboud, Nijmegen
  - UMC Utrecht, Utrecht